CLINICAL TRIAL: NCT03607422
Title: A Phase 3 Randomized, Placebo-Controlled, Double-Blind Study to Evaluate Upadacitinib in Adolescent and Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate Upadacitinib in Adolescents and Adults With Moderate to Severe Atopic Dermatitis (Measure Up 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M18-891; 2022-502936-38-00 (Other: EU CT)
Expanded Access: NCT04159597 (Available)
Record Dates: First submitted 2018-07-25; First posted 2018-07-31 (Actual); Results first posted 2022-03-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis; Upadacitinib; ABT-494; Measure Up 2
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo / Upadacitinib (Placebo Comparator): Participants will receive placebo orally once a day (QD) for 16 weeks in the double-blind treatment period. At Week 16 participants will be re-randomized to receive either upadacitinib 15 mg or upadacitinib 30 mg QD up to Week 260.
  Interventions: Drug: Placebo for Upadacitinib; Drug: Upadacitinib
- Upadacitinib 15 mg QD (Experimental): Participants will receive upadacitinib 15 mg orally once a day for up to 260 weeks.
  Interventions: Drug: Upadacitinib
- Upadacitinib 30 mg QD (Experimental): Participants will receive upadacitinib 30 mg orally once a day for up to 260 weeks.
  Interventions: Drug: Upadacitinib

INTERVENTIONS:
Drug: Placebo for Upadacitinib — Tablets taken orally once a day
  Arms: Placebo / Upadacitinib
Drug: Upadacitinib — Tablets taken orally once a day
  Other Names: ABT-494; RINVOQ®

SUMMARY:
The objective of this study is to assess the efficacy and safety of upadacitinib for the treatment of adolescent and adult participants with moderate to severe atopic dermatitis (AD) who are candidates for systemic therapy.

DETAILED DESCRIPTION:
This study includes a 35-day screening period, a 16-week double-blind period, a blinded extension period up to Week 260, and a 30-day follow-up visit.

Participants who meet eligibility criteria in the main study will be randomized in a 1:1:1 ratio to receive a daily oral dose of upadacitinib 30 mg or upadacitinib 15 mg or matching placebo. Upon completion of enrollment of a minimum of 810 participants in the main study, a supplemental study will continue to enroll adolescents (adolescent sub-study) until a total of 180 adolescent participants are enrolled overall (main study + adolescent sub-study).

Randomization in the main study will be stratified by baseline disease severity (validated Investigator Global Assessment scale for Atopic Dermatitis [vIGA-AD] score of moderate [3] versus severe [4]), by geographic region (United States [US]/Puerto Rico/Canada, and Other), and by age (adolescent [ages 12 to 17] versus adult [ages 18 to 75]). The separate randomization for the adolescent sub-study will be stratified by baseline disease severity (moderate [vIGA-AD = 3] vs. severe [vIGA-AD = 4]) and by geographic region (US/Puerto Rico/Canada and Other).

At Week 16 of the main study and the adolescent sub-study, participants in the placebo group will be re-randomized in a 1:1 ratio to receive daily oral doses of upadacitinib 30 mg or upadacitinib 15 mg in the blinded extension period. In the main study the re-randomization at Week 16 will be stratified by Week 16 50% improvement in Eczema Area and Severity Index [EASI 50] responder [Yes/No], geographic region [US/Puerto Rico/Canada, and other], and age group [adolescent/adult]. For the adolescent sub-study, the re-randomization will be stratified by EASI 50 responder (Yes/No) and by geographic region (US/Puerto Rico/Canada and Other). Participants originally randomized to upadacitinib will continue upadacitinib in the extension period at the same dose.

Starting at the Week 4 visit, rescue treatment for AD may be provided at the discretion of the investigator if medically necessary.

The Primary Analysis for the main study will be conducted after all ongoing participants have completed Week 16. In addition, a Primary Analysis for the adolescent population (including the adolescent participants from the main study and the adolescent sub-study) will be conducted after all ongoing adolescent participants have completed Week 16.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥ 40 kg at Baseline Visit for participants ≥ 12 and < 18 years of age
* Chronic atopic dermatitis (AD) with onset of symptoms at least 3 years prior to Baseline and subject meets Hanifin and Rajka criteria
* Active moderate to severe AD defined by Eczema Area and Severity Index (EASI) ≥ 16, validated Investigator's Global Assessment (vIGA) ≥ 3, body surface area (BSA) affected by AD ≥ 10%, and weekly average of daily Worst Pruritus numerical rating scale (NRS) score ≥ 4.
* Candidate for systemic therapy or have recently required systemic therapy for AD
* Documented history (within 6 months prior to Baseline) of inadequate response to topical corticosteroid (TCS) or topical calcineurin inhibitor (TCI) or documented systemic treatment for AD or for whom topical treatments are otherwise medically inadvisable due to side effects or safety risks

Exclusion Criteria:

* Prior exposure to any Janus kinase (JAK) inhibitor
* Unable or unwilling to discontinue current AD treatments prior to the study
* Requirement of prohibited medications during the study
* Other active skin diseases or skin infections requiring systemic treatment or would interfere with appropriate assessment of atopic dermatitis lesions
* Female subject who is pregnant, breastfeeding, or considering pregnancy during the study

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 912 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2025-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (196):
- United States (76):
  - Total Skin and Beauty Derm Ctr /ID# 205129, Birmingham, Alabama
  - Medical Dermatology Specialist /ID# 205516, Phoenix, Arizona
  - Arizona Research Center, Inc. /ID# 205795, Phoenix, Arizona
  - The Dermatology Clinic of Arkansas /ID# 218749, Bryant, Arkansas
  - Arkansas Research Trials /ID# 218469, North Little Rock, Arkansas
  - Encino Research Center /ID# 207472, Encino, California
  - University of California Irvine /ID# 205136, Irvine, California
  - Ark Clinical Research /ID# 218193, Long Beach, California
  - Keck School of Medicine of USC /ID# 206971, Los Angeles, California
  - Wallace Medical Group /ID# 205701, Los Angeles, California
  - Child Hosp of Orange County,CA /ID# 205735, Orange, California
  - Palmtree Clinical Research Inc. /Id# 206184, Palm Springs, California
  - Rady Children's Hospital San Diego /ID# 208244, San Diego, California
  - Southern California Derma. Inc /ID# 205734, Santa Ana, California
  - Innovative Clinical Research - Lafayette /ID# 208400, Lafayette, Colorado
  - New England Research Associates, LLC /ID# 206896, Bridgeport, Connecticut
  - Ideal Clinical Research Inc. /ID# 209880, Aventura, Florida
  - Skin Care Research, LLC /ID# 207099, Boca Raton, Florida
  - Midflorida Clinical Research, Inc. /ID# 213700, Brandon, Florida
  - Clinical Research of West Florida, Inc /ID# 206146, Clearwater, Florida
  - Revival Research /ID# 208383, Doral, Florida
  - Universal Axon Clinical Research /ID# 213703, Doral, Florida
  - Lakes Research, LLC /ID# 209156, Miami, Florida
  - Miami Dade Medical Research Institute /ID# 209413, Miami, Florida
  - Savin Medical Group, LLC /ID# 206902, Miami Lakes, Florida
  - Floridian Clinical Research /ID# 207433, Miami Lakes, Florida
  - Advanced Research for Health Improvement /ID# 217987, Naples, Florida
  - Advanced Research for Health Improvement /ID# 218003, Naples, Florida
  - Complete Health Research /ID# 213459, Ormond Beach, Florida
  - Precision Clinical Research /ID# 207364, Sunrise, Florida
  - Clinical Research Trials of Florida, Inc. /ID# 206840, Tampa, Florida
  - ForCare Clinical Research /ID# 205120, Tampa, Florida
  - Georgia Pollens Clinical Research Centers, Inc /ID# 218567, Albany, Georgia
  - Marietta Dermatology Clinical Research /ID# 210317, Marietta, Georgia
  - Agile Clinical Research Trials /ID# 218080, Sandy Springs, Georgia
  - Treasure Valley Medical Research /ID# 210298, Boise, Idaho
  - Great Lakes Clinical Trials /ID# 205830, Chicago, Illinois
  - Ashira Dermatology /ID# 205512, Gurnee, Illinois
  - Clinical Investigation Specialists, Inc. /ID# 206898, Gurnee, Illinois
  - Northshore University Health System Dermatology Clinical Trials Unit /ID# 205135, Skokie, Illinois
  - Raga Clinical Studies, LLC. /ID# 206749, Crown Point, Indiana
  - Hutchinson Clinic /ID# 205970, Hutchinson, Kansas
  - Continental Clinical Solutions /ID# 210327, Towson, Maryland
  - Beacon Clinical Research, LLC /ID# 206894, Quincy, Massachusetts
  - David Fivenson, MD, PLC /ID# 206903, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 206895, Ann Arbor, Michigan
  - Allergy, Asthma & Immunology Associates, PC /ID# 218169, Lincoln, Nebraska
  - Skin Specialists, PC /ID# 205515, Omaha, Nebraska
  - Duplicate_Summit Medical Group /ID# 213863, Clifton, New Jersey
  - Skin Laser and Surgery Specialists of NY and NJ /ID# 206754, Hackensack, New Jersey
  - Care Access Research /ID# 218476, Hoboken, New Jersey
  - University of New Mexico School of Medicine /ID# 206756, Albuquerque, New Mexico
  - Fordham Dermatology /ID# 218508, The Bronx, New York
  - PMG Research of Wilmington LLC /ID# 205968, Wilmington, North Carolina
  - University Hospitals Case Medical Center /ID# 206639, Cleveland, Ohio
  - Awasty Research Network, LLC /ID# 206748, Marion, Ohio
  - Southside Dermatology /ID# 214451, Tulsa, Oklahoma
  - Vital Prospects Clinical Research Institute, PC /ID# 205824, Tulsa, Oklahoma
  - Cyn3rgy Research /ID# 218064, Gresham, Oregon
  - Velocity Clinical Research Hallandale Beach /ID# 207544, Medford, Oregon
  - Clinical Research Solutions, LLC /ID# 218416, Jackson, Tennessee
  - Stones River Dermatology /ID# 205178, Murfreesboro, Tennessee
  - Metroplex Dermatology /ID# 213307, Arlington, Texas
  - Bellaire Dermatology /ID# 205470, Bellaire, Texas
  - Center for Clinical Studies /ID# 213186, Cypress, Texas
  - Dermatology Treatment and Research Center, PA /ID# 205473, Dallas, Texas
  - Epiphany Dermatology - Fort Worth /ID# 210073, Fort Worth, Texas
  - Styde Research, LLC /ID# 213469, Lewisville, Texas
  - Austin Institute for Clinical Research /ID# 206640, Pflugerville, Texas
  - Derm Clin Res Ctr San Antonio /ID# 205469, San Antonio, Texas
  - EPIC Medical Research /ID# 206382, Murray, Utah
  - Aspen Clinical Research /ID# 208399, Orem, Utah
  - Timber Lane Allergy & Asthma Research, LLC /ID# 206897, South Burlington, Vermont
  - The Education & Research Foundation, Inc. /ID# 206900, Lynchburg, Virginia
  - Bellingham Asthma Allergy and Immunology Clinic /ID# 210357, Bellingham, Washington
  - Clinical Investigation Specialist, Inc - Kenosha /ID# 215933, Kenosha, Wisconsin
- Australia (7):
  - The Skin Hospital /ID# 217846, Westmead, New South Wales
  - The Skin Centre /ID# 205922, Benowa, Queensland
  - Box Hill Hospital /ID# 206023, Box Hill, Victoria
  - Monash Children's Hospital /ID# 217917, Clayton, Victoria
  - Sinclair Dermatology /ID# 217791, East Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 205919, Parkville, Victoria
  - Murdoch Children's Research Institute /ID# 205667, Parkville, Victoria
- Austria (4):
  - Universitaetsklinikum St. Poelten /ID# 206909, Sankt Pölten, Lower Austria
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 206573, Linz, Upper Austria
  - Klinik Donaustadt /ID# 206572, Vienna, Vienna
  - Landeskrankenhaus Salzburg-Universitätsklinikum der PMU (LKH) /ID# 208281, Salzburg
- Belgium (3):
  - UCL Saint-Luc /ID# 205537, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent /ID# 205181, Ghent, Oost-Vlaanderen
  - Centre Hospitalier Universitaire du Sart Tilman CHU de Liege /ID# 204938, Liège
- Bulgaria (4):
  - Medical center Sveti Panteleimon /ID# 210414, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 205292, Sofia
  - Military Medical Academy Multiprofile Hospital /ID# 205291, Sofia
  - Medical complex Doverie /ID# 211289, Sofia
- Canada (15):
  - Stratica Medical /ID# 205415, Edmonton, Alberta
  - Alberta DermaSurgery Centre /ID# 205422, Edmonton, Alberta
  - UBC Department of Dermatology and Skin Science The Skin Care Centre /ID# 207837, Vancouver, British Columbia
  - Pacific Derm /ID# 206797, Vancouver, British Columbia
  - Skin Care Studio /ID# 205420, St. John's, Newfoundland and Labrador
  - SimcoDerm Medical and Surgical Dermatology Center /ID# 206333, Barrie, Ontario
  - Kingsway Clinical Research /ID# 206005, Etobicoke, Ontario
  - Dr. Lyne Giroux Medicine Professional Corporation /ID# 206771, Greater Sudbury, Ontario
  - Dr. Dusan Sajic Medicine Professional Corporation /ID# 206890, Guelph, Ontario
  - The Guenther Dermatology Research Centre /ID# 206772, London, Ontario
  - DermEdge Research Inc. /ID# 206036, Mississauga, Ontario
  - Dr. S.K. Siddha Medicine Professional Corporation /ID# 207138, Newmarket, Ontario
  - Allergy Research Canada Inc. /ID# 213547, Niagara Falls, Ontario
  - Niakosari Medicine Professional Corporation /ID# 206004, Toronto, Ontario
  - Skinsense Medical Research /ID# 206873, Saskatoon, Saskatchewan
- Croatia (4):
  - DermaPlus - Poliklinika za dermatologiju i venerologiju /ID# 205429, Zagreb, City of Zagreb
  - Djecja bolnica Srebrnjak /ID# 205926, Zagreb, City of Zagreb
  - Poliklinika Vlatka Cavka d.o.o. /ID# 211126, Zagreb, City of Zagreb
  - Naftalan - Specijalna bolnica za medicinsku rehabilitaciju /ID# 203448, Ivanić-Grad, Zagreb County
- Czechia (5):
  - Fakultni nemocnice Plzen /ID# 205096, Pilsen
  - Sanatorium profesora Arenbergera /ID# 205098, Prague
  - Vseobecna fakultni nemocnice v Praze /ID# 205201, Prague
  - Fakultni Nemocnice v Motole /ID# 218192, Prague
  - Krajska zdravotni, a.s. - Masarykova nemocnice v Usti nad Labem, o. z. /ID# 205097, Ústí nad Labem
- Denmark (2):
  - Aarhus University Hospital /ID# 205524, Aarhus N, Central Jutland
  - Sjællands Universitetshospital /ID# 205960, Roskilde, Region Sjælland
- France (5):
  - Hopital Saint-Andre /ID# 206554, Bordeaux
  - CHRU de Brest - Hopital Morvan /ID# 206555, Brest
  - C.H. de Bretagne Sud /ID# 206910, Lorient
  - AP-HP - Hopital Saint-Louis /ID# 206552, Paris
  - Hopital Prive d'Antony /ID# 206553, Antony, Île-de-France Region
- Germany (8):
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 206658, Kiel, Schleswig-Holstein
  - Klinikum Darmstadt /ID# 207483, Darmstadt
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 205767, Dresden
  - Universitaetsklinikum Hamburg-Eppendorf (UKE) /ID# 207982, Hamburg
  - Dermatologische Gemeinschaftspraxis Mahlow /ID# 205765, Mahlow
  - Haut- und Laserzentrum Hunsrück /ID# 205768, Simmern
  - Hautarztpraxis Dr. med. Matthias Hoffmann /ID# 205766, Witten
  - CentroDerm GmbH /ID# 206861, Wuppertal
- Greece (4):
  - 251 Airforce General Hospital /ID# 205841, Athens, Attica
  - 401 GSNA - 401 Army General Hospital /ID# 205352, Athens, Attica
  - General Hospital Andreas Syggros /ID# 204527, Athens, Attica
  - Papageorgiou General Hospital Thessaloniki /ID# 204526, Stavroupoli (Thessalonikis), Thessaloniki
- Hungary (7):
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz /ID# 218072, Miskolc, Borsod-Abauj Zemplen county
  - Bugat Pal Korhaz /ID# 211247, Gyöngyös, Heves County
  - Somogy Megyei Kaposi Mor Oktato Korhaz /ID# 205611, Kaposvár, Somogy County
  - Drug Research Center /ID# 217855, Balatonfüred, Veszprém megye
  - Clinexpert Kft /ID# 211246, Budapest
  - Synexus Magyarorszag Kft. /ID# 206008, Budapest
  - Pecsi Tudomanyegyetem Klinikai Kozpont /ID# 205085, Pécs
- Ireland (4):
  - St James Hospital /ID# 204264, Dublin, Dublin
  - South Infirmary Victoria University Hospital /ID# 204265, Cork
  - University Hospital Galway /ID# 209965, Galway
  - University Hospital Waterford /ID# 204266, Waterford
- Italy (6):
  - IRCCS Istituti Fisioterapici Ospitalieri-Istituto Dermatologico San Gallicano /ID# 205986, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 205987, Rome, Lazio
  - ASST Spedali civili di Brescia /ID# 205927, Brescia
  - Azienda Ospedaliero Universitaria di Cagliari- Presidio Ospedaliero /ID# 205168, Cagliari
  - Presidio Ospedaliero San Salvatore /ID# 205167, L’Aquila
  - Azienda Ospedaliero-Universitaria di Modena /ID# 205169, Modena
- Netherlands (4):
  - Bravis Ziekenhuis /ID# 206676, Bergen op Zoom, North Brabant
  - Centrum Oosterwal /ID# 209640, Alkmaar
  - Reinier de Graaf /ID# 205811, Delft
  - Universitair Medisch Centrum Groningen /ID# 205162, Groningen
- Greenlane Clinical Centre /ID# 205664, Epsom, Auckland, New Zealand
- Portugal (6):
  - CCA Braga - Hospital de Braga /ID# 205854, Braga
  - Centro Hospitalar de Leiria, EPE /ID# 209906, Leiria
  - Centro Hospitalar Universitário de Lisboa Norte, EPE - Hospital de Santa Maria /ID# 205839, Lisbon
  - Hospital CUF Descobertas /ID# 205431, Lisbon
  - CHP, EPE- Hospital Geral de Sa /ID# 205187, Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE /ID# 205679, Porto
- Singapore (5):
  - National Skin Centre /ID# 205222, Singapore, Central Singapore
  - National University Hospital /ID# 205224, Singapore
  - Singapore General Hospital /ID# 205225, Singapore
  - KK Women's & Children Hospital /ID# 206693, Singapore
  - Changi General Hospital /ID# 205223, Singapore
- South Korea (7):
  - Korea University Ansan Hospital /ID# 206342, Ansan, Gyeonggido
  - SoonChunHyang University Buchon Hospital /ID# 206391, Habun, Gyeonggido
  - Ajou University Hospital /ID# 206341, Suwon, Gyeonggido
  - The Catholic University of Korea Incheon St.Mary's Hospital /ID# 206529, Incheon
  - Seoul National University Hospital /ID# 206396, Seoul
  - Chung-Ang University Hostipal /ID# 206397, Seoul
  - Hallym University Kangnam Sacred Heart Hospital /ID# 206343, Seoul
- Spain (10):
  - Hospital Sant Joan de Deu /ID# 218047, Esplugues de Llobregat, Barcelona
  - Hospital Vital Alvarez Buylla /ID# 205770, Mieres, Principality of Asturias
  - Hospital Parc de Salut del Mar /ID# 204709, Barcelona
  - Hospital Clinic de Barcelona /ID# 210564, Barcelona
  - Hospital Universitario Reina Sofia /ID# 204712, Córdoba
  - Hospital Campus de la Salud /ID# 205544, Granada
  - Hospital General Universitario Gregorio Maranon /ID# 204380, Madrid
  - Hospital Infantil Universitario Nino Jesus /ID# 210437, Madrid
  - Hospital Universitario Infanta Leonor /ID# 204710, Madrid
  - Hospital General Universitario de Valencia /ID# 210565, Valencia
- Taiwan (4):
  - Taipei Medical University Shuang Ho Hospital /ID# 204804, New Taipei City
  - Chung Shan Medical University Hospital /ID# 205092, Taichung
  - National Taiwan University Hospital /ID# 204803, Taipei
  - Linkou Chang Gung Memorial Ho /ID# 204783, Taoyuan
- United Kingdom (5):
  - University Hospital Southampton NHS Foundation Trust /ID# 205711, Southampton, Hampshire
  - Northwick Park Hospital /ID# 205250, Middlesex, Harrow
  - Barts Health NHS Trust /ID# 206491, London, London, City of
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 204993, Newcastle upon Tyne
  - University Hospital Plymouth NHS Trust /ID# 204649, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Irvine AD, Prajapati VH, Guttman-Yassky E, Simpson EL, Papp KA, Blauvelt A, Chu CY, Hong HC, Gold LFS, de Bruin-Weller M, Bieber T, Kabashima K, Rosmarin D, Sancho C, Calimlim BM, Grada A, Yang Y, Wu X, Levy G, Raymundo EM, Teixeira HD, Silverberg JI. Efficacy and Safety of Upadacitinib in Patients With Moderate-to-Severe Atopic Dermatitis: Phase 3 Randomized Clinical Trial Results Through 140 Weeks. Am J Clin Dermatol. 2025 Nov;26(6):1003-1016. doi: 10.1007/s40257-025-00975-3. Epub 2025 Sep 3. PMID 40900410
- [Derived] Burmester GR, Deodhar A, Irvine AD, Panaccione R, Winthrop KL, Vleugels RA, Levy G, Suravaram S, Palac H, Wegrzyn L, Ford S, Meerwein S, Guttman-Yassky E. Safety Profile of Upadacitinib: Descriptive Analysis in Over 27,000 Patient-Years Across Rheumatoid Arthritis, Psoriatic Arthritis, Axial Spondyloarthritis, Atopic Dermatitis, and Inflammatory Bowel Disease. Adv Ther. 2025 Oct;42(10):5215-5237. doi: 10.1007/s12325-025-03328-y. Epub 2025 Aug 28. PMID 40875187
- [Derived] Silverberg JI, Gooderham M, Katoh N, Aoki V, Pink AE, Binamer Y, Glick B, Staubach P, Calimlim B, Li C, Grada A, Moreira A, Lee WJ, Wollenberg A. Achieving Optimal Treatment Targets and Minimal Disease Activity with Upadacitinib for Moderate-to-Severe Atopic Dermatitis: Integrated Analysis of Phase 3 Studies (Measure Up 1 and 2). Dermatol Ther (Heidelb). 2025 Sep;15(9):2583-2594. doi: 10.1007/s13555-025-01485-0. Epub 2025 Jul 14. PMID 40658277
- [Derived] Simpson EL, Silverberg JI, Prajapati VH, Eyerich K, Katoh N, Boguniewicz M, Guttman-Yassky E, Song EJ, Lee WJ, Teixeira HD, Wu T, Sancho Sanchez C, Vigna N, Calimlim BM, de Bruin-Weller M. Rapid Itch Improvement and Skin Clearance with Upadacitinib Versus Placebo (Measure Up 1 and Measure Up 2) and Versus Dupilumab (Heads Up): Results from Three Phase 3 Clinical Trials in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Aug;15(8):2061-2076. doi: 10.1007/s13555-025-01443-w. Epub 2025 Jun 2. PMID 40457140
- [Derived] Paller AS, Mendes-Bastos P, Siegfried E, Eichenfield LF, Soong W, Prajapati VH, Lio P, Simpson EL, Raymundo EM, Suravaram S, Hu X, Yang Y, Huang X, Calimlim BM, Platt AM, Su JC, Zheng M, Yamamoto-Hanada K, Teixeira HD, Irvine AD. Upadacitinib in Adolescents With Moderate to Severe Atopic Dermatitis: Analysis of 3 Phase 3 Randomized Clinical Trials Through 76 Weeks. JAMA Dermatol. 2024 Dec 1;160(12):1304-1313. doi: 10.1001/jamadermatol.2024.3696. PMID 39441580
- [Derived] Blauvelt A, Eyerich K, Irvine AD, de Bruin-Weller M, Kwatra SG, Gooderham M, Kim B, Calimlim BM, Lee WJ, Raymundo EM, Liu Y, Ofori S, Platt AM, Silverberg JI. More Time Spent with Clear Skin and No Itch with Upadacitinib versus Dupilumab for Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2621-2630. doi: 10.1007/s13555-024-01242-9. Epub 2024 Aug 7. PMID 39110139
- [Derived] Simpson EL, Prajapati VH, Leshem YA, Chovatiya R, de Bruin-Weller MS, Stander S, Pink AE, Calimlim BM, Lee WJ, Teixeira H, Ladizinski B, Hu X, Yang Y, Liu Y, Liu M, Grada A, Platt AM, Silverberg JI. Upadacitinib Rapidly Improves Patient-Reported Outcomes in Atopic Dermatitis: 16-Week Results from Phase 3 Clinical Trials (Measure Up 1 and 2). Dermatol Ther (Heidelb). 2024 May;14(5):1127-1144. doi: 10.1007/s13555-024-01157-5. Epub 2024 May 2. PMID 38696027
- [Derived] Silverberg JI, Gooderham MJ, Paller AS, Deleuran M, Bunick CG, Gold LFS, Hijnen D, Calimlim BM, Lee WJ, Teixeira HD, Hu X, Zhang S, Yang Y, Grada A, Platt AM, Thaci D. Early and Sustained Improvements in Symptoms and Quality of Life with Upadacitinib in Adults and Adolescents with Moderate-to-Severe Atopic Dermatitis: 52-Week Results from Two Phase III Randomized Clinical Trials (Measure Up 1 and Measure Up 2). Am J Clin Dermatol. 2024 May;25(3):485-496. doi: 10.1007/s40257-024-00853-4. Epub 2024 Mar 25. PMID 38528257
- [Derived] Thyssen JP, Thaci D, Bieber T, Gooderham M, de Bruin-Weller M, Soong W, Kabashima K, Barbarot S, Luna PC, Xu J, Hu X, Liu Y, Raymundo EM, Calimlim BM, Nduaka C, Gamelli A, Simpson EL. Upadacitinib for moderate-to-severe atopic dermatitis: Stratified analysis from three randomized phase 3 trials by key baseline characteristics. J Eur Acad Dermatol Venereol. 2023 Sep;37(9):1871-1880. doi: 10.1111/jdv.19232. Epub 2023 Jun 21. PMID 37247226
- [Derived] Paller AS, Ladizinski B, Mendes-Bastos P, Siegfried E, Soong W, Prajapati VH, Lio P, Thyssen JP, Simpson EL, Platt AM, Raymundo EM, Liu J, Calimlim BM, Huang X, Gu Y, Hu X, Yang Y, Su JC, Zheng M, Yamamoto-Hanada K, Teixeira HD, Irvine AD. Efficacy and Safety of Upadacitinib Treatment in Adolescents With Moderate-to-Severe Atopic Dermatitis: Analysis of the Measure Up 1, Measure Up 2, and AD Up Randomized Clinical Trials. JAMA Dermatol. 2023 May 1;159(5):526-535. doi: 10.1001/jamadermatol.2023.0391. PMID 37043227
- [Derived] Burmester GR, Cohen SB, Winthrop KL, Nash P, Irvine AD, Deodhar A, Mysler E, Tanaka Y, Liu J, Lacerda AP, Palac H, Shaw T, Mease PJ, Guttman-Yassky E. Safety profile of upadacitinib over 15 000 patient-years across rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis and atopic dermatitis. RMD Open. 2023 Feb;9(1):e002735. doi: 10.1136/rmdopen-2022-002735. PMID 36754548
- [Derived] Mendes-Bastos P, Ladizinski B, Guttman-Yassky E, Jiang P, Liu J, Prajapati VH, Simpson EL, Vigna N, Teixeira HD, Barbarot S. Characterization of acne associated with upadacitinib treatment in patients with moderate-to-severe atopic dermatitis: A post hoc integrated analysis of 3 phase 3 randomized, double-blind, placebo-controlled trials. J Am Acad Dermatol. 2022 Oct;87(4):784-791. doi: 10.1016/j.jaad.2022.06.012. Epub 2022 Jun 15. PMID 35714786
- [Derived] Simpson EL, Papp KA, Blauvelt A, Chu CY, Hong HC, Katoh N, Calimlim BM, Thyssen JP, Chiou AS, Bissonnette R, Stein Gold LF, Wegzyn C, Hu X, Liu M, Liu J, Tenorio AR, Chu AD, Guttman-Yassky E. Efficacy and Safety of Upadacitinib in Patients With Moderate to Severe Atopic Dermatitis: Analysis of Follow-up Data From the Measure Up 1 and Measure Up 2 Randomized Clinical Trials. JAMA Dermatol. 2022 Apr 1;158(4):404-413. doi: 10.1001/jamadermatol.2022.0029. PMID 35262646
- [Derived] Guttman-Yassky E, Teixeira HD, Simpson EL, Papp KA, Pangan AL, Blauvelt A, Thaci D, Chu CY, Hong HC, Katoh N, Paller AS, Calimlim B, Gu Y, Hu X, Liu M, Yang Y, Liu J, Tenorio AR, Chu AD, Irvine AD. Once-daily upadacitinib versus placebo in adolescents and adults with moderate-to-severe atopic dermatitis (Measure Up 1 and Measure Up 2): results from two replicate double-blind, randomised controlled phase 3 trials. Lancet. 2021 Jun 5;397(10290):2151-2168. doi: 10.1016/S0140-6736(21)00588-2. Epub 2021 May 21. PMID 34023008
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 154 study sites in 23 countries across Europe, North America, Oceania, and the Asia-Pacific region.
  The study included a 16-week double-blind treatment period followed by an ongoing blinded extension period.
  The first 836 adults and adolescents enrolled constituted the Main Study; additional adolescents were enrolled in the Adolescent Substudy to ensure enrollment of a total of 180 adolescent participants overall.
  Results are reported up to Week 16.
Pre-assignment Details: Participants were randomized equally into 1 of 3 treatment groups, stratified by disease severity (validated Investigator Global Assessment Scale for Atopic Dermatitis [vIGA-AD] moderate [3] vs severe [4]), geographic region (US/Puerto Rico/Canada vs Other), and age (adolescent [ages 12 to 17] vs adult [ages 18 to 75]). Randomization for the adolescent substudy was stratified by disease severity (vIGA-AD 3 vs vIGA-AD 4) and geographic region (US/Puerto Rico/Canada vs Other).
Groups:
- Adults: Placebo: Participants ≥ 18 years old received placebo orally once a day (QD) for 16 weeks.
- Adults: Upadacitinib 15 mg QD: Participants ≥ 18 years old received upadacitinib 15 mg orally once a day for 16 weeks.
- Adults: Upadacitinib 30 mg QD: Participants ≥ 18 years old received upadacitinib 30 mg orally once a day for 16 weeks.
- Adolescents: Placebo: Adolescent participants (12 - 17 years old) received placebo orally once a day for 16 weeks.
- Adolescents: Upadacitinib 15 mg QD: Adolescent participants received upadacitinib 15 mg orally once a day for 16 weeks.
- Adolescents: Upadacitinib 30 mg QD: Adolescent participants received upadacitinib 30 mg orally once a day for 16 weeks.
Period: Overall Study
Arm/Group | Adults: Placebo | Adults: Upadacitinib 15 mg QD | Adults: Upadacitinib 30 mg QD | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Started (Randomized into study) | 242 | 243 | 247 | 60 | 58 | 62
Completed (Completed Week 16) | 204 | 233 | 235 | 55 | 55 | 59
Not Completed | 38 | 10 | 12 | 5 | 3 | 3
Not completed — Adverse Event | 7 | 3 | 2 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 11 | 3 | 6 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other | 12 | 4 | 1 | 2 | 0 | 2
Not completed — Ongoing at Time of Analysis | 8 | 0 | 2 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Adults: Placebo: Participants ≥ 18 years old received placebo orally once a day for 16 weeks.
- Adolescents: Placebo: Adolescent participants received placebo orally once a day for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Adults: Placebo | Adults: Upadacitinib 15 mg QD | Adults: Upadacitinib 30 mg QD | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD | Total
Number analyzed (Participants) | 242 | 243 | 247 | 60 | 58 | 62 | 912
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (14.08) | 35.7 (15.15) | 36.7 (15.36) | 15.5 (1.67) | 15.2 (1.79) | 15.8 (1.70) | 32.1 (15.66)
Age, Customized [Count of Participants; unit: Participants]
  12 - 14 years | 0 | 0 | 0 | 18 | 23 | 15 | 56
  15 - 17 years | 0 | 0 | 0 | 42 | 35 | 47 | 124
  18 - < 40 years | 161 | 165 | 161 | 0 | 0 | 0 | 487
  40 - < 65 years | 70 | 63 | 67 | 0 | 0 | 0 | 200
  ≥ 65 years | 11 | 15 | 19 | 0 | 0 | 0 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 102 | 103 | 35 | 38 | 26 | 408
  Male | 138 | 141 | 144 | 25 | 20 | 36 | 504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 18 | 17 | 10 | 12 | 11 | 93
  Not Hispanic or Latino | 217 | 225 | 230 | 50 | 46 | 51 | 819
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 1 | 0 | 2 | 1 | 13
  Asian | 52 | 62 | 55 | 6 | 5 | 12 | 192
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2 | 0 | 4
  Black or African American | 15 | 16 | 17 | 7 | 5 | 3 | 63
  White | 165 | 160 | 172 | 45 | 42 | 46 | 630
  More than one race | 4 | 1 | 2 | 1 | 2 | 0 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Study Enrollment [Count of Participants; unit: Participants]
  Main Study | 242 | 243 | 247 | 36 | 33 | 35 | 836
  Adolescent Substudy | 0 | 0 | 0 | 24 | 25 | 27 | 76
Geographic Region [Count of Participants; unit: Participants]
  US/Puerto Rico/Canada | 95 | 95 | 99 | 25 | 24 | 27 | 365
  Other | 147 | 148 | 148 | 35 | 34 | 35 | 547
vIGA-AD [Count of Participants; unit: Participants] — The vIGA-AD was used to assess the severity of AD based on lesion appearance on the following scale:
  * 0-Clear: No inflammatory signs of AD;
  * 1-Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  * 2-Mild: Slight but definite erythema, induration/papulation and/or lichenification. No oozing or crusting;
  * 3-Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4-Severe: Marked erythema, induration/papulation and/or lichenification, oozing or crusting may be present.
  Participants
    3 (Moderate) | 110 | 111 | 111 | 26 | 27 | 29 | 414
    4 (Severe) | 132 | 132 | 136 | 34 | 31 | 33 | 498
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: score on a scale] — EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease. Population: Participants with available data
  score on a scale
    number analyzed (Participants) | 241 | 243 | 247 | 60 | 58 | 62 | 911
    (all) | 28.74 (11.865) | 28.65 (11.633) | 29.61 (12.030) | 30.12 (13.263) | 28.01 (12.216) | 31.15 (13.998) | 29.16 (12.112)
Disease Duration since Diagnosis [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 242 | 243 | 246 | 60 | 58 | 62 | 911
    (all) | 22.263 (14.0798) | 19.802 (13.8089) | 21.911 (14.8401) | 12.169 (4.7104) | 11.184 (4.5479) | 12.128 (4.6414) | 19.452 (13.4892)

OUTCOME MEASURES:

1. Primary Outcome: Main Study: Percentage of Participants Achieving at Least a 75% Reduction in Eczema Area and Severity Index Score (EASI 75) From Baseline at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/ neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: The intent-to-treat population for the main study (ITT_M) includes all participants who were randomized in the main study (adults and adolescents). Non-responder imputation incorporating multiple imputation to handle missing data due to coronavirus disease 2019 pandemic (COVID-19) (NRI-C) was used.
  The pre-specified primary analysis included participants enrolled in the main study only; Efficacy analyses of adolescent participants were conducted separately and are reported below.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo: Participants received placebo orally once a day for 16 weeks.
- Upadacitinib 15 mg QD: Participants received upadacitinib 15 mg orally once a day for 16 weeks.
- Upadacitinib 30 mg QD: Participants received upadacitinib 30 mg orally once a day for 16 weeks.
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 278 | 276 | 282
percentage of participants | 13.3 [9.3 to 17.3] | 60.1 [54.4 to 65.9] | 72.9 [67.7 to 78.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 30 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 59.6, 95% CI 2-sided [53.1 to 66.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 15 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 46.9, 95% CI 2-sided [39.9 to 53.9] — Response Rate Difference = Upadacitinib - Placebo

2. Primary Outcome: Main Study: Percentage of Participants Achieving Validated Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) of 0 or 1 With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No inflammatory signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification, no oozing or crusting;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification, no oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 278 | 276 | 282
percentage of participants | 4.7 [2.2 to 7.2] | 38.8 [33.0 to 44.5] | 52.0 [46.1 to 57.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 47.4, 95% CI 2-sided [41.0 to 53.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 34.0, 95% CI 2-sided [27.8 to 40.2] — Response Rate Difference = Upadacitinib - Placebo

3. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus Numerical Rating Scale (NRS) at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Worst Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with Worst Pruritus NRS (weekly average) ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 274 | 270 | 280
percentage of participants | 9.1 [5.7 to 12.5] | 41.9 [36.0 to 47.7] | 59.6 [53.9 to 65.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 50.4, 95% CI 2-sided [43.8 to 57.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 32.6, 95% CI 2-sided [25.8 to 39.4] — Response Rate Difference = Upadacitinib - Placebo

4. Secondary Outcome: Main Study: Percentage of Participants Achieving a 90% Reduction From Baseline in EASI Score (EASI 90) at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 278 | 276 | 282
percentage of participants | 5.4 [2.7 to 8.1] | 42.4 [36.6 to 48.2] | 58.5 [52.7 to 64.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 53.1, 95% CI 2-sided [46.7 to 59.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 36.9, 95% CI 2-sided [30.6 to 43.3] — Response Rate Difference = Upadacitinib - Placebo

5. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 4
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 274 | 270 | 280
percentage of participants | 3.6 [1.4 to 5.9] | 48.9 [42.9 to 54.9] | 60.7 [55.0 to 66.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 57.0, 95% CI 2-sided [50.9 to 63.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 45.2, 95% CI 2-sided [38.9 to 51.4] — Response Rate Difference = Upadacitinib - Placebo

6. Secondary Outcome: Main Study: Percentage of Participants Achieving an EASI 75 Response at Week 2
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 75 response is defined as at least a 75% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 278 | 276 | 282
percentage of participants | 3.6 [1.4 to 5.8] | 33.0 [27.4 to 38.5] | 44.0 [38.2 to 49.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 40.4, 95% CI 2-sided [34.2 to 46.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 29.4, 95% CI 2-sided [23.5 to 35.3] — Response Rate Difference = Upadacitinib - Placebo

7. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 1
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 274 | 270 | 280
percentage of participants | 0.7 [0.0 to 1.7] | 7.4 [4.3 to 10.5] | 15.7 [11.5 to 20.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 14.9, 95% CI 2-sided [10.6 to 19.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 6.7, 95% CI 2-sided [3.4 to 10.0] — Response Rate Difference = Upadacitinib - Placebo

8. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 2
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11- point scale from 0 (no itch) to 10 (worst imaginable itch). The percentage of participants who had a 4-point or greater improvement from Baseline in Worst Pruritus NRS score at Day 2 was pre-specified as a ranked secondary endpoint for participants in the upadacitinib 30 mg group versus placebo group only.
Time Frame: Baseline and Day 2
Population: Intent-to-treat population for the main study with Worst Pruritus NRS (daily score) ≥ 4 at Baseline; Non-responder imputation with no special data handling for missing data due to COVID-19 (NRI-NC) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 267 | 269 | 278
percentage of participants | 0.7 [0.0 to 1.8] | 7.4 [4.3 to 10.6] | 7.9 [4.7 to 11.1]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 7.2, 95% CI 2-sided [3.8 to 10.5] — Response Rate Difference = Upadacitinib - Placebo

9. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 3
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
  The percentage of participants who had a 4-point or greater improvement in Worst Pruritus NRS score from Baseline at Day 3 was pre-specified as a ranked secondary endpoint for participants in the upadacitinib 15 mg group versus placebo group only.
Time Frame: Baseline and Day 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 267 | 269 | 278
percentage of participants | 3.0 [1.0 to 5.0] | 11.5 [7.7 to 15.3] | 17.3 [12.8 to 21.7]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 8.6, 95% CI 2-sided [4.3 to 12.9] — Response Rate Difference = Upadacitinib - Placebo

10. Secondary Outcome: Main Study: Percentage of Participants Experiencing a Flare During the Double-blind Treatment Period
Description: A flare, characterized as a clinically meaningful worsening in EASI, is defined as an increase in EASI score of ≥ 6.6 points from Baseline during the double-blind treatment period and prior to use of any rescue medication. Flare was assessed in participants with an EASI score of 65.4 or less at Baseline.
Time Frame: From first dose of study drug to Week 16
Population: Intent-to-treat population for the main study with an EASI score ≤ 65.4 at Baseline and at least one EASI post-baseline assessment prior to use of rescue medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 269 | 274 | 277
percentage of participants | 24.5 [19.4 to 29.7] | 2.2 [0.5 to 3.9] | 1.4 [0.0 to 2.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = -23.1, 95% CI 2-sided [-28.4 to -17.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = -22.4, 95% CI 2-sided [-27.8 to -16.9] — Response Rate Difference = Upadacitinib - Placebo

11. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 12 Points From Baseline in Atopic Dermatitis Impact Scale (ADerm-IS) Sleep Domain Score at Week 16
Description: The ADerm-IS is a 10-item patient reported outcome (PRO) questionnaire designed to assess a variety of impacts that participants experience from their AD.
  The ADerm-IS sleep domain consists of 3 questions designed to assess the impact of AD on sleep on a daily basis over a 24-hour recall period. The items include difficulty falling asleep, impact on sleep, and waking at night. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The ADerm-IS sleep domain score is the sum of the 3 item scores and ranges from 0 (no impact) to 30 (worst impact). The ADerm-IS sleep domain was analyzed based on weekly rolling averages of daily scores.
  The minimal clinically important difference for ADerm-IS sleep domain score is 12.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with ADerm-IS Sleep Domain score ≥ 12 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 233 | 219 | 228
percentage of participants | 12.4 [8.2 to 16.7] | 50.2 [43.6 to 56.9] | 62.3 [56.0 to 68.6]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 49.8, 95% CI 2-sided [42.2 to 57.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 37.9, 95% CI 2-sided [30.1 to 45.8] — Response Rate Difference = Upadacitinib - Placebo

12. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Atopic Dermatitis Symptom Scale (ADerm-SS) Skin Pain Score at Week 16
Description: The ADerm-SS is an 11-item PRO questionnaire designed to assess signs and symptoms that patients may experience due to AD using a 24-hour recall period. For the skin pain item participants were asked on a daily basis to indicate how bad their worst skin pain due to AD was in the past 24 hours on an NRS from 0 (no pain) to 10 (worst imaginable pain). The ADerm-SS skin pain score was analyzed using weekly rolling averages of daily scores. The minimal clinically important difference for ADerm-SS skin pain score is 4.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with ADerm-SS Skin Pain Score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 247 | 237 | 238
percentage of participants | 13.4 [9.1 to 17.6] | 49.4 [43.0 to 55.7] | 65.1 [59.1 to 71.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 51.8, 95% CI 2-sided [44.4 to 59.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 35.9, 95% CI 2-sided [28.2 to 43.5] — Response Rate Difference = Upadacitinib - Placebo

13. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 28 Points From Baseline in ADerm-SS 7-Item Total Symptom Score (TSS-7) at Week 16
Description: The ADerm-SS is an 11-item questionnaire designed to assess signs and symptoms that participants may experience due to AD using a 24-hour recall period. The 7-item total symptom score includes 7 symptoms (items 1-7 of the ADerm-SS), each assessed on a NRS from 0 (no symptom) to 10 (worst imaginable). The 7 symptoms included in the score are itch while asleep, itch while awake, skin pain (each assessed daily), skin cracking, skin cracking pain, dry skin, and skin flaking (assessed weekly). The TSS-7 score ranges from 0 to 70, with higher scores indicating worsening symptoms. The minimal clinically important difference for ADerm-SS TSS-7 is 28.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with ADerm-SS TSS-7 ≥ 28 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 244 | 230 | 234
percentage of participants | 12.7 [8.5 to 16.9] | 53.0 [46.6 to 59.5] | 66.2 [60.2 to 72.3]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 53.3, 95% CI 2-sided [46.0 to 60.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 40.3, 95% CI 2-sided [32.7 to 48.0] — Response Rate Difference = Upadacitinib - Placebo

14. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 11 Points From Baseline in ADerm-IS Emotional State Domain Score at Week 16
Description: The ADerm-IS is a 10-item PRO questionnaire designed to assess a variety of impacts that participants experience from their AD.
  ADerm-IS emotional state sums three items [Items 8-10] measuring self-consciousness, embarrassment, and sadness with a 7-day recall. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The emotional state domain score ranges from 0 to 30, where higher scores represent worst impact.
  The minimal clinically important difference for ADerm-IS emotional state domain score is 11.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with ADerm-IS Emotional State domain score ≥ 11 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 234 | 228 | 228
percentage of participants | 16.7 [11.9 to 21.4] | 57.0 [50.6 to 63.4] | 71.5 [65.6 to 77.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 54.8, 95% CI 2-sided [47.2 to 62.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 40.3, 95% CI 2-sided [32.3 to 48.3] — Response Rate Difference = Upadacitinib - Placebo

15. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 14 Points From Baseline in ADerm-IS Daily Activities Domain Score at Week 16
Description: The ADerm-IS is a 10-item PRO questionnaire designed to assess a variety of impacts that participants experience from their AD.
  ADerm-IS Daily Activities sums four items measuring limitations of household, physical, and social activities, and difficulty concentrating with a 7-day recall. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The daily activities domain score ranges from 0 to 40, where higher scores represent worst impact.
  The minimal clinically important difference for the ADerm-IS daily activities domain score is 14.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with ADerm-IS Daily Activities Domain Score ≥ 14 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 227 | 207 | 223
percentage of participants | 18.9 [13.8 to 24.0] | 57.0 [50.3 to 63.7] | 69.5 [63.5 to 75.5]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 50.6, 95% CI 2-sided [42.8 to 58.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 37.9, 95% CI 2-sided [29.5 to 46.3] — Response Rate Difference = Upadacitinib - Placebo

16. Secondary Outcome: Main Study: Percentage of Participants Achieving a 100% Reduction From Baseline in EASI Score (EASI 100) at Week 16
Description: as for outcome 4
Time Frame: Baseline and Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 278 | 276 | 282
percentage of participants | 0.7 [0.0 to 1.7] | 14.1 [10.0 to 18.2] | 18.8 [14.2 to 23.4]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 18.1, 95% CI 2-sided [13.5 to 22.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 1, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 13.4, 95% CI 2-sided [9.2 to 17.6] — Response Rate Difference = Upadacitinib - Placebo

17. Secondary Outcome: Main Study: Percent Change From Baseline in Worst Pruritus NRS at Week 16
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Worst Pruritus NRS was analyzed based on weekly rolling averages of daily scores. A negative change from Baseline indicates improvement.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for the main study with non-missing Baseline and Week 16 values; missing data were handled using a mixed-effect model with repeated measurements (MMRM) including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 119 | 224 | 235
percent change | -17.04 [-22.39 to -11.69] | -51.20 [-55.80 to -46.61] | -66.49 [-71.03 to -61.96]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 30 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for European Union (EU)/European Medicines Agency (EMA) regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, Baseline vIGA-AD category and age in the model; Least Squares (LS) Mean Difference = -49.45, 95% CI 2-sided [-56.05 to -42.84], Standard Error of Mean 3.364 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 15 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -34.16, 95% CI 2-sided [-40.81 to -27.51], Standard Error of Mean 3.386 — Difference = Upadacitinib - Placebo

18. Secondary Outcome: Main Study: Percent Change From Baseline in EASI Score at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1)] moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 142 | 246 | 250
percent change | -34.51 [-39.60 to -29.42] | -74.13 [-78.45 to -69.82] | -84.65 [-88.93 to -80.37]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — The overall type I error rate of the primary and secondary endpoints for upadacitinib 30 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -50.14, 95% CI 2-sided [-56.28 to -44.00], Standard Error of Mean 3.127 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -39.62, 95% CI 2-sided [-45.79 to -33.46], Standard Error of Mean 3.139 — Difference = Upadacitinib - Placebo

19. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Patient Oriented Eczema Measure (POEM) Total Score at Week 16
Description: The POEM is a 7-item, validated questionnaire used to assess disease symptoms in both children and adults.
  Participants respond to 7 questions, including dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping, each scored on a 5-point scale based on frequency of occurrence during the previous week: 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days. Item scores are added to provide a total score ranging from 0 (clear) to 28 (very severe atopic eczema). A change in POEM score of 3.4 points is considered the minimal clinically important difference.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study with POEM score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 268 | 268 | 269
percentage of participants | 28.7 [23.3 to 34.1] | 70.9 [65.5 to 76.3] | 83.5 [79.1 to 88.0]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 54.7, 95% CI 2-sided [47.7 to 61.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; The overall type I error rate of the primary and secondary endpoints for upadacitinib 15 mg was strongly controlled using a graphical multiple testing procedure at the two-sided 0.05 level following a pre-specified α transfer path which includes downstream transfer along the endpoints sequence within each dose as well as cross-dose transfer. This endpoint was a multiplicity-controlled key secondary endpoint for EU/EMA regulatory purposes only; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 42.1, 95% CI 2-sided [34.5 to 49.8] — Response Rate Difference = Upadacitinib - Placebo

20. Secondary Outcome: Main Study: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL.
  the DLQI was administered to participants who were ≥ 16 (16 to 75) years old at the time of the Screening visit.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for the main study who were ≥ 16 years old at Screening with DLQI score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 250 | 251 | 251
percentage of participants | 28.4 [22.8 to 34.0] | 71.7 [66.1 to 77.3] | 77.6 [72.5 to 82.8]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 49.0, 95% CI 2-sided [41.4 to 56.5] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p = 0.002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 42.8, 95% CI 2-sided [35.0 to 50.6] — Response Rate Difference = Upadacitinib - Placebo

21. Secondary Outcome: Main Study: Percent Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score at Week 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: as for outcome 17
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 136 | 245 | 241
percent change | -28.43 [-33.34 to -23.52] | -57.90 [-61.84 to -53.97] | -68.44 [-72.44 to -64.44]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -40.01, 95% CI 2-sided [-45.80 to -34.22], Standard Error of Mean 2.949 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 17, analysis 1]; LS Mean Difference = -29.47, 95% CI 2-sided [-35.24 to -23.69], Standard Error of Mean 2.941

22. Secondary Outcome: Main Study: Percentage of Participants Achieving a Hospital Anxiety and Depression Scale-Anxiety (HADS-A) Score and Hospital Anxiety and Depression Scale-Depression (HADS-D) Score of < 8 at Week 16
Description: The HADS is a 14-item questionnaire, with seven items related to anxiety (HADS-A) and seven items related to depression (HADS-D). Each item is scored from 0 to 3; scores for each subscale range from 0 to 21, with higher scores indicating more distress. For each domain, scores 7 or lower are considered normal, 8 to 10 are borderline, and 11 or higher indicate clinical anxiety or depression.
Time Frame: Week 16
Population: Intent-to-treat population for the main study with HADS-A ≥ 8 or HADS-D ≥ 8 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 140 | 137 | 146
percentage of participants | 11.4 [6.2 to 16.7] | 46.0 [37.6 to 54.3] | 56.1 [48.1 to 64.2]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 44.5, 95% CI 2-sided [35.0 to 54.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 34.4, 95% CI 2-sided [24.7 to 44.2] — Response Rate Difference = Upadacitinib - Placebo

23. Secondary Outcome: Main Study: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 16
Description: The DLQI is a 10-item validated questionnaire used to assess the impact of AD disease symptoms and treatment on quality of life (QoL). It consists of 10 questions evaluating impact of skin diseases on different aspects of a participant's QoL over the prior week, including symptoms and feelings, daily activities, leisure, work or school, personal relationships, and the side effects of treatment. Each item is scored on a 4-point scale (0 = not at all/not relevant; 1 = a little; 2 = a lot; and 3 = very much).
  Item scores are added to provide a total score, ranging from 0 to 30, with higher scores indicating greater impairment of QoL. A score of 0 or 1 means that the disease has no effect at all.
  The DLQI was administered to participants who were ≥ 16 (16 to 75) years old at the time of the Screening visit.
Time Frame: Week 16
Population: Intent-to-treat population for the main study who were ≥ 16 years old at Screening with DLQI score > 1 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 15 mg QD | Upadacitinib 30 mg QD
Number analyzed (Participants) | 257 | 252 | 256
percentage of participants | 4.7 [2.1 to 7.2] | 23.8 [18.6 to 29.1] | 37.9 [32.0 to 43.9]
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg QD; Test type: Superiority — [test comment as in outcome 18, analysis 1]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 33.3, 95% CI 2-sided [26.9 to 39.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg QD; Test type: Superiority — [test comment as in outcome 17, analysis 2]; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for strata (Baseline vIGA-AD categories and age [adolescent vs. adult]); Adjusted Response Rate Difference = 19.1, 95% CI 2-sided [13.3 to 24.9] — Response Rate Difference = Upadacitinib - Placebo

24. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 16
Description: as for outcome 6
Time Frame: Baseline and Week 16
Population: The ITT population for adolescents (ITT_A) consists of all adolescent participants who were randomized in the main study or the adolescent sub-study. Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 58 | 62
percentage of participants | 13.3 [4.7 to 21.9] | 69.0 [57.1 to 80.9] | 73.4 [62.3 to 84.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 59.9, 95% CI 2-sided [45.9 to 73.8] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 55.8, 95% CI 2-sided [41.1 to 70.4] — Response Rate Difference = Upadacitinib - Placebo

25. Secondary Outcome: Adolescents: Percentage of Participants Achieving a vIGA-AD of 0 or 1 With a Reduction From Baseline of ≥ 2 Points at Week 16
Description: The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification, no oozing or crusting;;
  * 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification, no oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; possible oozing or crusting.
Time Frame: Baseline and Week 16
Population: The ITT population for adolescents; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 58 | 62
percentage of participants | 5.0 [0.0 to 10.5] | 44.8 [32.0 to 57.6] | 59.4 [47.0 to 71.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 53.9, 95% CI 2-sided [40.6 to 67.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 39.4, 95% CI 2-sided [25.7 to 53.1] — Response Rate Difference = Upadacitinib - Placebo

26. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 16
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with Worst Pruritus NRS (weekly average) ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 55 | 60
percentage of participants | 3.4 [0.0 to 8.0] | 38.2 [25.3 to 51.0] | 56.7 [44.1 to 69.2]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 53.1, 95% CI 2-sided [40.0 to 66.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 35.0, 95% CI 2-sided [21.8 to 48.2] — Response Rate Difference = Upadacitinib - Placebo

27. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 90 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 90 response is defined as at least a 90% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 58 | 62
percentage of participants | 1.7 [0.0 to 4.9] | 48.3 [35.4 to 61.1] | 62.0 [49.8 to 74.3]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 60.2, 95% CI 2-sided [47.5 to 72.9] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 46.7, 95% CI 2-sided [33.4 to 59.9] — Response Rate Difference = Upadacitinib - Placebo

28. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 4
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 4
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 55 | 60
percentage of participants | 3.4 [0.0 to 8.0] | 38.2 [25.3 to 51.0] | 50.0 [37.3 to 62.7]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 46.4, 95% CI 2-sided [33.2 to 59.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 34.9, 95% CI 2-sided [21.4 to 48.4] — Response Rate Difference = Upadacitinib - Placebo

29. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 75 Response at Week 2
Description: as for outcome 6
Time Frame: Baseline and Week 2
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 58 | 62
percentage of participants | 6.7 [0.4 to 13.0] | 37.9 [25.4 to 50.4] | 53.2 [40.8 to 65.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 46.2, 95% CI 2-sided [32.4 to 60.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 31.3, 95% CI 2-sided [17.3 to 45.3] — Response Rate Difference = Upadacitinib - Placebo

30. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Week 1
Description: as for outcome 3
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 1
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 55 | 60
percentage of participants | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 12.7 [3.9 to 21.5] | 5.0 [0.0 to 10.5]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p = 0.075, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 5.0, 95% CI 2-sided [-0.5 to 10.6] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.005, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 12.7, 95% CI 2-sided [3.9 to 21.5] — Response Rate Difference = Upadacitinib - Placebo

31. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 2
Description: Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch).
Time Frame: Baseline and Day 2
Population: Intent-to-treat population for adolescents with Worst Pruritus NRS (daily score) ≥ 4 at Baseline; Non-responder imputation with no special data handling for missing data due to COVID-19 was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 56 | 62
percentage of participants | 0.0 [NA to NA] — Could not be calculated using the normal approximation to the binomial distribution | 8.9 [1.5 to 16.4] | 3.2 [0.0 to 7.6]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p = 0.151, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 3.2, 95% CI 2-sided [-1.2 to 7.6] — Response Rate Difference = Upadacitinib - Placebo

32. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in Worst Pruritus NRS at Day 3
Description: as for outcome 31
Time Frame: Baseline and Day 3
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 59 | 56 | 62
percentage of participants | 1.7 [0.0 to 5.0] | 14.3 [5.1 to 23.5] | 9.7 [2.3 to 17.0]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 12.9, 95% CI 2-sided [3.4 to 22.3] — Response Rate Difference = Upadacitinib - Placebo

33. Secondary Outcome: Adolescents: Percentage of Participants Experiencing a Flare During the Double-blind Treatment Period
Description: A flare, characterized as a clinically meaningful worsening in EASI, is defined as an increase in EASI score of ≥ 6.6 points from Baseline during the double-blind treatment period and prior to use of any rescue medication. Flares were assessed in participants with an EASI score of 65.4 or less at Baseline.
Time Frame: From first dose of study drug to Week 16
Population: Intent-to-treat population for adolescents with an EASI score ≤ 65.4 at Baseline and at least one EASI post-baseline assessment prior to use of rescue medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 58 | 61
percentage of participants | 20.0 [9.9 to 30.1] | 1.7 [0.0 to 5.1] | 1.6 [0.0 to 4.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = -18.0, 95% CI 2-sided [-28.0 to -8.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = -17.9, 95% CI 2-sided [-28.1 to -7.7] — Response Rate Difference = Upadacitinib - Placebo

34. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 12 Points From Baseline in ADerm-IS Sleep Domain Score at Week 16
Description: The ADerm-IS is a 10-item patient reported outcome questionnaire designed to assess a variety of impacts that participants experience from their AD.
  The ADerm-IS sleep domain consists of 3 questions designed to assess the impact of AD on sleep on a daily basis over a 24-hour recall period. The items include difficulty falling asleep, impact on sleep, and waking at night. Each question is scored on an 11-point NRS from 0 (no impact) to 10 (extreme impact). The ADerm-IS sleep domain score is the sum of the 3 item scores and ranges from 0 (no impact) to 30 (worst impact). The ADerm-IS sleep domain was analyzed based on weekly rolling averages of daily scores.
  The minimal clinically important difference for ADerm-IS sleep domain score is 12.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with ADerm-IS Sleep Domain score ≥ 12 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 42 | 40 | 44
percentage of participants | 9.5 [0.6 to 18.4] | 37.5 [22.5 to 52.5] | 61.4 [47.0 to 75.8]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 51.5, 95% CI 2-sided [34.8 to 68.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 29.2, 95% CI 2-sided [11.8 to 46.6] — Response Rate Difference = Upadacitinib - Placebo

35. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in ADerm-SS Skin Pain Score at Week 16
Description: The ADerm-SS is an 11-item PRO questionnaire designed to assess signs and symptoms that patients may experience due to AD using a 24-hour recall period. For the skin pain item participants were asked to indicate on a daily basis how bad their worst skin pain due to AD was in the past 24 hours on an NRS from 0 (no pain) to 10 (worst imaginable pain).
  The minimal clinically important difference for ADerm-SS skin pain score is 4. The ADerm-SS skin pain score was analyzed based on weekly rolling averages of daily scores.
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with ADerm-SS Skin Pain score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 53 | 48 | 51
percentage of participants | 7.5 [0.4 to 14.7] | 39.6 [25.7 to 53.4] | 60.8 [47.4 to 74.2]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 53.2, 95% CI 2-sided [38.4 to 68.0] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 31.8, 95% CI 2-sided [16.5 to 47.1] — Response Rate Difference = Upadacitinib - Placebo

36. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 28 Points From Baseline in ADerm-SS TSS-7 at Week 16
Description: as for outcome 13
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with ADerm-SS TSS-7 ≥ 28 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 55 | 48 | 55
percentage of participants | 10.9 [2.7 to 19.1] | 47.9 [33.8 to 62.0] | 60.0 [47.1 to 72.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 48.9, 95% CI 2-sided [33.8 to 64.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 37.3, 95% CI 2-sided [21.1 to 53.6] — Response Rate Difference = Upadacitinib - Placebo

37. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 11 Points From Baseline in ADerm-IS Emotional State Domain Score at Week 16
Description: as for outcome 14
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with ADerm-IS Emotional State Domain score ≥ 11 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 50 | 45 | 50
percentage of participants | 18.0 [7.4 to 28.6] | 60.0 [45.7 to 74.3] | 72.0 [59.6 to 84.4]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 53.8, 95% CI 2-sided [37.4 to 70.2] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 42.0, 95% CI 2-sided [24.3 to 59.7] — Response Rate Difference = Upadacitinib - Placebo

38. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 14 Points From Baseline in ADerm-IS Daily Activities Domain Score at Week 16
Description: as for outcome 15
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with ADerm-IS Daily Activities Domain Score ≥ 14 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 49 | 40 | 50
percentage of participants | 22.4 [10.8 to 34.1] | 52.5 [37.0 to 68.0] | 68.0 [55.1 to 80.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 45.3, 95% CI 2-sided [28.0 to 62.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 29.8, 95% CI 2-sided [10.7 to 48.8] — Response Rate Difference = Upadacitinib - Placebo

39. Secondary Outcome: Adolescents: Percentage of Participants Achieving an EASI 100 Response at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 100 response is defined as a 100% reduction (improvement) from Baseline in EASI score.
Time Frame: Baseline and Week 16
Population: as for outcome 25
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 60 | 58 | 62
percentage of participants | 1.7 [0.0 to 4.9] | 15.5 [6.2 to 24.8] | 19.4 [9.5 to 29.2]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 17.1, 95% CI 2-sided [7.5 to 26.7] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 13.7, 95% CI 2-sided [3.9 to 23.5] — Response Rate Difference = Upadacitinib - Placebo

40. Secondary Outcome: Adolescents: Percent Change From Baseline in Worst Pruritus NRS at Week 16
Description: as for outcome 17
Time Frame: Baseline (last available rolling average before the first dose of study drug) and Week 16
Population: Intent-to-treat population for adolescents with non-missing Baseline and Week 16 values; missing data were handled using a mixed-effect model with repeated measurements including observed measurements at all visits, except that measurements after any rescue medication were excluded.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 27 | 49 | 55
percent change | -11.02 [-22.14 to 0.10] | -47.56 [-57.00 to -38.13] | -66.95 [-76.07 to -57.84]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, and Baseline vIGA-AD category in the model; LS Mean Difference = -55.93, 95% CI 2-sided [-70.32 to -41.55], Standard Error of Mean 7.284 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 40, analysis 1]; LS Mean Difference = -36.54, 95% CI 2-sided [-51.12 to -21.96], Standard Error of Mean 7.384 — Difference = Upadacitinib - Placebo

41. Secondary Outcome: Adolescents: Percent Change From Baseline in EASI Score at Week 16
Description: as for outcome 18
Time Frame: Baseline and Week 16
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 31 | 53 | 52
percent change | -42.19 [-52.06 to -32.33] | -77.85 [-85.95 to -69.74] | -84.81 [-92.84 to -76.78]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 40, analysis 1]; LS Mean Difference = -42.62, 95% CI 2-sided [-55.34 to -29.90], Standard Error of Mean 6.432 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 40, analysis 1]; LS Mean Difference = -35.66, 95% CI 2-sided [-48.41 to -22.90], Standard Error of Mean 6.447 — Difference = Upadacitinib - Placebo

42. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in POEM Total Score at Week 16
Description: as for outcome 19
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents with POEM score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 57 | 56 | 57
percentage of participants | 28.1 [16.4 to 39.7] | 66.1 [53.7 to 78.5] | 80.7 [70.5 to 90.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 52.5, 95% CI 2-sided [36.9 to 68.1] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 38.1, 95% CI 2-sided [21.2 to 54.9] — Response Rate Difference = Upadacitinib - Placebo

43. Secondary Outcome: Adolescents: Percentage of Participants Achieving a Reduction of ≥ 4 Points From Baseline in DLQI Score at Week 16
Description: as for outcome 20
Time Frame: Baseline and Week 16
Population: Intent-to-treat population for adolescents who were ≥ 16 years old at Screening with DLQI score ≥ 4 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 26 | 22 | 30
percentage of participants | 19.2 [4.1 to 34.4] | 68.2 [48.7 to 87.6] | 73.3 [57.5 to 89.2]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 55.9, 95% CI 2-sided [35.5 to 76.3] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 49.6, 95% CI 2-sided [26.3 to 72.9] — Response Rate Difference = Upadacitinib - Placebo

44. Secondary Outcome: Adolescents: Percent Change From Baseline in SCORAD Score at Week 16
Description: as for outcome 21
Time Frame: Baseline and Week 16
Population: as for outcome 40
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 30 | 54 | 49
percent change | -27.91 [-37.98 to -17.83] | -57.89 [-65.49 to -50.28] | -72.81 [-80.77 to -64.85]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; Mixed-effect model repeat measurement with Baseline, treatment, visit, treatment by visit interaction, and Baseline vIGA-AD category; LS Mean Difference = -44.90, 95% CI 2-sided [-57.74 to -32.06], Standard Error of Mean 6.492 — Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p < 0.001, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 44, analysis 1]; LS Mean Difference = -29.98, 95% CI 2-sided [-42.60 to -17.36], Standard Error of Mean 6.383 — Difference = Upadacitinib - Placebo

45. Secondary Outcome: Adolescents: Percentage of Participants Achieving HADS-A Score and HADS-D Score of < 8 at Week 16
Description: as for outcome 22
Time Frame: Week 16
Population: Intent-to-treat population for adolescents with HADS-A ≥ 8 or HADS-D ≥ 8 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 25 | 24 | 32
percentage of participants | 16.0 [1.6 to 30.4] | 37.5 [18.1 to 56.9] | 43.8 [26.6 to 60.9]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p = 0.016, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 27.8, 95% CI 2-sided [5.2 to 50.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.062, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 22.3, 95% CI 2-sided [-1.1 to 45.7] — Response Rate Difference = Upadacitinib - Placebo

46. Secondary Outcome: Adolescents: Percentage of Participants Achieving a DLQI Score of 0 or 1 at Week 16
Description: as for outcome 23
Time Frame: Week 16
Population: Intent-to-treat population for adolescents who were ≥ 16 years old at Screening with DLQI score > 1 at Baseline; Non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C) was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
Number analyzed (Participants) | 26 | 22 | 32
percentage of participants | 7.7 [0.0 to 17.9] | 13.6 [0.0 to 28.0] | 46.9 [29.6 to 64.2]
Statistical Analysis 1: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 30 mg QD; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 38.9, 95% CI 2-sided [18.4 to 59.4] — Response Rate Difference = Upadacitinib - Placebo
Statistical Analysis 2: Comparison: Adolescents: Placebo vs Adolescents: Upadacitinib 15 mg QD; Test type: Superiority; p = 0.510, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (Baseline vIGA-AD categories); Adjusted Response Rate Difference = 5.9, 95% CI 2-sided [-11.7 to 23.6] — Response Rate Difference = Upadacitinib - Placebo

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 16, or 30 days after last dose for participants who did not enter the blinded extension period.
Arm/Group | Adults: Placebo | Adults: Upadacitinib 15 mg QD | Adults: Upadacitinib 30 mg QD | Adolescents: Placebo | Adolescents: Upadacitinib 15 mg QD | Adolescents: Upadacitinib 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/242 | 0/243 | 0/247 | 0/60 | 0/58 | 0/62
Serious Adverse Events (participants affected / at risk) | 6/242 | 3/243 | 7/247 | 3/60 | 2/58 | 0/62
Other Adverse Events (participants affected / at risk) | 52/242 | 78/243 | 94/247 | 15/60 | 21/58 | 25/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults: Placebo (N=242) | Adults: Upadacitinib 15 mg QD (N=243) | Adults: Upadacitinib 30 mg QD (N=247) | Adolescents: Placebo (N=60) | Adolescents: Upadacitinib 15 mg QD (N=58) | Adolescents: Upadacitinib 30 mg QD (N=62)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL TEAR (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECZEMA HERPETICUM (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IMPETIGO (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEAT STROKE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
PNEUMOMEDIASTINUM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults: Placebo (N=242) | Adults: Upadacitinib 15 mg QD (N=243) | Adults: Upadacitinib 30 mg QD (N=247) | Adolescents: Placebo (N=60) | Adolescents: Upadacitinib 15 mg QD (N=58) | Adolescents: Upadacitinib 30 mg QD (N=62)
FATIGUE (General disorders) | 2 (2) | 2 (2) | 8 (9) | 0 (0) | 3 (3) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 11 (20) | 14 (17) | 18 (18) | 2 (2) | 2 (2) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (13) | 13 (14) | 14 (19) | 1 (1) | 6 (6) | 3 (3)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 4 (5) | 8 (8) | 10 (10) | 1 (1) | 3 (3) | 6 (6)
HEADACHE (Nervous system disorders) | 10 (11) | 17 (20) | 16 (17) | 2 (4) | 3 (4) | 5 (6)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (5) | 2 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 4 (5) | 0 (0) | 4 (4) | 2 (2)
ACNE (Skin and subcutaneous tissue disorders) | 5 (5) | 31 (32) | 38 (39) | 2 (2) | 6 (6) | 9 (10)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 17 (19) | 7 (7) | 2 (2) | 8 (8) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT03607422/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT03607422/SAP_001.pdf